CLINICAL TRIAL: NCT01506869
Title: A Prospective Cohort Study on the Associations of Diabetes With Cancer Risk in Chinese Men and Women
Brief Title: Risk Evaluation of cAncers in Chinese diabeTic Individuals: a lONgitudinal Study
Acronym: REACTION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Chinese Society of Endocrinology (Unknown)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Other Study IDs: CCEMD010
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples were collected and retained for biomarker analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Type 2 diabetes
- Prediabetes
- Normal glucose regulation

SUMMARY:
Phase 1: Baseline investigation (nation-wide survey)

Aims: To investigate whether diabetes and prediabetes is a risk factor for cancers of all sites as well as for specific type of cancer, such as breast and colorectal cancer.

Subjects and Methods: A nation-wide survey will be carried out in 200,000-250,000 individuals selected from 20-25 communities stratified according to geographic regions (northeast, north, east, south central, northwest, and southwest China), degrees of urbanization (large cities [Beijing, Shanghai, and provincial capitals], midsize cities, county seats, and rural townships), and economic development status (as assessed on the basis of the gross domestic product [GDP] for each province). A comprehensive examination including questionnaire, anthropometric measurements, biochemical analysis will be performed in each study participant. Diabetes and prediabetes should be diagnosed by OGTT according to the WHO 1999 criteria, while the diagnosis of cancer is established on the self-report questionnaire and cross checking with the tumor registry or a proof of doctor's diagnosis.

Phase 2: Cohort follow-up

Aims : To examine factors that modify the risk of cancer in diabetes, prediabetes and normal glucose regulation (NGR).

Subjects and Methods: To recruit and follow all type 2 diabetes, prediabetes, and sex,age-matched NGR (1:1) in each community for at least 3 years. For diabetes, treatment target is HbA1c ≤ 7.0% with treatment paradigm recommended by local guideline.

ELIGIBILITY:
Phase 1

Inclusion Criteria:

1. Age >= 40 years old
2. Gender: males and females
3. Provide written informed consent
4. Satisfactory compliance

Phase 2

Inclusion Criteria:

1. Age >= 40 and =< 75 years old
2. Gender: males and females
3. Provide written informed consent
4. Satisfactory compliance

Exclusion Criteria:

1. History of cancer;
2. History of LADA and other autoimmunity diseases;
3. Acute diabetic complication, acidosis, etc;
4. Moderate to severe liver, kidney dysfunction, i.e. ALT/AST > 2.5 times the upper limit of normal range or Ccr < 25ml/min;
5. Any other condition or major systemic diseases that the investigator feels would interfere with trial participation or evaluation of results.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In phase 1, 200,000-250,000 individuals selected from 20-25 communities stratified according to geographic regions, degrees of urbanization, and economic development status In Phase 2, 30,000-40,000 type 2 diabetes, 20,000-30,000 prediabetes, 30,000-40,000 normal glucose regulation, recruited from the baseline survey
Sampling Method: Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
number of participants who develop cancer during follow-up | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD,PHD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao-Tong University School of Medicine, Shanghai, China

REFERENCES:
- [Derived] Wang L, Wu P, Chen K, Li B, Wang J, Mu Y. Correlation between rate-pressure product or pressure-rate quotient and urinary albumin-creatinine ratio in the Chinese older population: The REACTION study. Chin Med J (Engl). 2024 Jan 20;137(2):238-240. doi: 10.1097/CM9.0000000000002941. Epub 2024 Jan 8. No abstract available. PMID 38185831
- [Derived] Xu C, Zhou G, Zhao M, Zhang X, Fang L, Guan Q, Zhang H, Gao L, Zhang T, Zhao J. Bidirectional temporal relationship between obesity and hyperinsulinemia: longitudinal observation from a Chinese cohort. BMJ Open Diabetes Res Care. 2021 Feb;9(1):e002059. doi: 10.1136/bmjdrc-2020-002059. PMID 33632707
- [Derived] Chen Y, Lin H, Qin L, Lu Y, Zhao L, Xia M, Jiang J, Li X, Yu C, Zong G, Zheng Y, Gao X, Su Q, Li X. Fasting Serum Fructose Levels Are Associated With Risk of Incident Type 2 Diabetes in Middle-Aged and Older Chinese Population. Diabetes Care. 2020 Sep;43(9):2217-2225. doi: 10.2337/dc19-2494. Epub 2020 Jul 1. PMID 32611608